CLINICAL TRIAL: NCT04108533
Title: LATcH: Lactation Achievement With Texts at Home
Brief Title: Lactation Achievement With Texts at Home
Acronym: LATcH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Celeste Durnwald, Principal Investigator, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 833824
Record Dates: First submitted 2019-09-25; First posted 2019-09-30 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Breastfeeding; Breastfeeding, Exclusive; Postpartum Depression
MeSH Terms: conditions — Breast Feeding; Depression, Postpartum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Text-Based Support (Experimental): Text-Based Support - Women randomized to this arm will receive text-based support via the Way to Health platform as described below.
  Supportive texts - Encouraging text messages with prompts to ask questions will be sent twice weekly during the first four weeks postpartum and once weekly thereafter for the remaining two weeks of the program
  Inquiry texts - Questions regarding infant feeding with prompts to answer will be sent three times weekly during the first two weeks postpartum and twice weekly thereafter for the remaining 4 weeks of the program.
  PHQ2 text - Women will be sent the PHQ2 at 2 weeks and 6 weeks postpartum to assess mood symptoms.
  Women in this group will also have the option to send a text with a question or concern at any time during the study. Weekdays from 8am to 5 pm these will be fielded by a trained obstetrician. If a text is received after-hours or on the weekend, women will be instructed to reach out to their primary OBGYN provider.
  Interventions: Behavioral: Text-Based Support
- Usual Care (No Intervention): Usual care - Women randomized to this arm will receive usual postpartum care with the following exceptions:
  Inquiry texts- Questions regarding infant feeding with prompts to answer will be sent once weekly for all 6 weeks of the program.
  PHQ2 text - Women will be sent the PHQ2 at 2 weeks and 6 weeks postpartum to assess mood symptoms.
  Women in this group will be directed to their physician with any questions or concerns during the study period.

INTERVENTIONS:
Behavioral: Text-Based Support — Text-based breastfeeding support as described in arm/group descriptions
  Arms: Text-Based Support

SUMMARY:
The objective of this study is to determine if text-based breastfeeding support improves breastfeeding initiation, exclusivity, and duration when compared to usual postpartum care. All women without a contraindication to breastfeeding and access to a mobile phone with unlimited text messaging capability who deliver a healthy term neonate will be eligible for inclusion. Consented women will be randomized to either text-based breastfeeding support using the Way to Health platform or usual care.

DETAILED DESCRIPTION:
Breastfeeding is a public health priority. The CDC and WHO, among other professional organizations, have issued the following recommendations with respect to breastmilk. Infants should be exclusively breastfed through the first 6 months of life and continue to receive breastmilk through at least the first year of life. Many women, however, are not meeting these benchmarks even among those who desire to do so. Approximately one quarter of infants are exclusively breastfed at 6 months and a little over 1/3 are still receiving breastmilk at the time of their 1st birthday.1 What looking at these numbers alone miss is the number of women who attempt to breastfeed and do not continue to do so. 83% of women attempt breastfeeding indicating that there is a significant drop off that occurs between delivery and 6 and 12 months of life.

While the risk factors for this are vast, lack of education poor socioeconomic status and poor social support are important contributors to breastfeeding problems. Both professional and informal support through family or friends have a significant impact on breastfeeding outcomes. Not all patients, however, have the resources needed to obtain professional support or the family experience necessary to meet their breastfeeding goals.

Digital support in other medical specialties have shown success in health outcomes. Multiple international studies have also demonstrated the benefits of text-messaging on breastfeeding rates including improved rates and duration of exclusivity. Thus far, none of these studies have been performed in the United States.

Therefore, the aim of this study is to determine if text-based breastfeeding support improves breastfeeding initiation, duration, and exclusivity when compared to usual postpartum care.

All women without a contraindication to breastfeeding and access to a mobile phone with unlimited text messaging capability will be approached in the 34-36 week of pregnancy.

All consented women will be enrolled in a "run-in" period in which they receive weekly text messages with factual information about breastfeeding. A response is required to one or more of these texts in order to be eligible for randomization at delivery.

Upon delivery of a healthy term neonate, women who responded in the "run-in" period will be randomized to either text-based breastfeeding support using the Way to Health platform or usual care.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* English-speaking
* Own a cellular phone with unlimited text-messaging
* Singleton gestation consented at 34-36 weeks of pregnancy
* Willing and able to sign consent form

Exclusion Criteria:

* Contraindication to breastfeeding
* Delivery of infant requiring ICN admission
* Physician discretion that patient will be unable to comply with the protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Exclusivity | 6 weeks postpartum
  Exclusive breastfeeding

SECONDARY OUTCOMES:
Any Breastfeeding | 6 weeks postpartum
  Any reported breastfeeding
Duration | 6 weeks postpartum
  Duration of breastfeeding
Formula | 6 weeks postpartum
  Rate of formula use
Compliance | 6 weeks postpartum
  Compliance with postpartum visit
Mood | 2 and 6 weeks postpartum
  Mood assessment using PHQ-2

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of the University Of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bender W, Levine L, Durnwald C. Text Message-Based Breastfeeding Support Compared With Usual Care: A Randomized Controlled Trial. Obstet Gynecol. 2022 Nov 1;140(5):853-860. doi: 10.1097/AOG.0000000000004961. Epub 2022 Oct 5. PMID 36201773